CLINICAL TRIAL: NCT05215873
Title: Oxytocin Versus Oral Misoprostol for Induction of Labor in Pregnant Women With Term Prelabor Rupture of Membranes
Brief Title: Induction of Labor in Pregnant Women With Prelabor Rupture of Membranes - Oxytocin or Misoprostol
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Rania Hassan Mostafa, Principal Investigator, Ain Shams Maternity Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMASU MS 733/2020/2021
Record Dates: First submitted 2022-01-05; First posted 2022-01-31 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Prelabor Rupture of Membranes
Keywords: oxytocin; misoprostol
MeSH Terms: conditions — Fetal Membranes, Premature Rupture | interventions — Misoprostol; Oxytocin

STUDY DESIGN:
Intervention Model Description: * 1st group (misoprostol group): induction of labor by 25µg misoprostol oral tablet every 4 hours with maximum200 µg.
  * 2nd group (oxytocin group:control group): induction of labor done by administration of oxytocin infusion according to ASUMH local protocol.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- misoprostol group (Active Comparator): 25µg misoprostol oral tablet every 4 hours with maximum200 µg
  Interventions: Drug: Misoprostol
- oxytocin group (Active Comparator): oxytocin infusion according to ASUMH local protocol: Put 3IU oxytocin (3000mIU) +50ml of normal saline in syringe pump= (60mIU/ml). Commence at 1ml/hour (1mIU/min) for 1/2 hour.
  * If contractions inadequate +fetal monitor healthy 2 ml/hour for 1/2 hour.
  * If contractions inadequate +fetal monitor healthy 4 ml/hour for 1/2 hour.
  * If contractions inadequate +fetal monitor healthy 6 ml/hour for 1/2 hour.
  * If contractions inadequate +fetal monitor healthy increase by 2ml/hr. for max. 27ml/hour.
  At any point there's fetal or maternal distress (e.g. pathological FHR pattern, antepartum hemorrhage, etc.) the study intervention will be stopped, and the maternal/fetal condition will be managed by cesarean section.
  Interventions: Drug: Syntocinon

INTERVENTIONS:
Drug: Misoprostol — a synthetic prostaglandin E1 analogue
  Other Names: vagiprost
  Arms: misoprostol group
Drug: Syntocinon — synthetic oxytocin
  Other Names: oxytocin
  Arms: oxytocin group

SUMMARY:
The aim of study is to compare the efficacy and safety of oral misoprostol versus oxytocin in induction of labor in pregnant women with prelabor rupture of membranes at term.

DETAILED DESCRIPTION:
Type of Study: Randomized controlled clinical trial. Study Setting: The study will be conducted at Ain Shams University Maternity Hospital (ASUMH) at labor ward.

Study Population: pregnant women attending at Ain Shams University Maternity Hospital for induction of labor at term

Sample Size: The study will be conducted on (170) women; they will be subdivided into 2 groups.

* 1st group (misoprostol group): induction of labor by 25µg misoprostol oral tablet every 4 hours with maximum200 µg.
* 2nd group (oxytocin group:control group): induction of labor done by administration of oxytocin infusion according to ASUMH local protocol.
* Sample size Justification: Using PASS 11program for sample size calculation and according to (Zeteroğlu S et al, 2006), the expected mean interval from induction to delivery in misoprostol group=10.61 ± 2.45 hours and oxytocin group=11.57 ± 1.91 hours. Sample size of 85 women per group can detect the difference between two group with power80% setting alpha error at 0.05.

Study procedures and interventions:

1. After approval of study protocol; pregnant women attending Ain Shams University Maternity Hospital for induction of labor will be enrolled into the study according to inclusion and exclusion criteria.
2. History taking, examination and investigation will be done to choose eligible patients.

   History: personal, obstetric history, past history (any medical or surgical disorder)

   Examination:

   General: pulse, blood pressure, temperature. Abdominal: size of the uterus, previous scar, presentation Per vaginal examination (PV): assessment of Bishop Score. Investigations: Routine laboratory: (CBC, Urine analysis, blood group and Rh typing) and ultrasound for (viability of fetus, fetal biometry and estimated fetal weight, amniotic fluid, placental localization), admission fetal heart rate (FHR) assessment (non-stress test "NST")
3. Eligible patients will be randomized using a computer-generated sequence 1:1 either to the misoprostol group or to oxytocin group.

The supervisor will do all procedures. Randomization: Will be done using computer generated randomization sheet using Med calc. ©.

Allocation and concealment: will be done using sealed opaque envelopes. Each woman will be invited to pull out an envelope, and according to the letter within she will be allocated to either group (group A: oral misoprostol; group B: oxytocin group) 4. Intervention:

1. st group (Misoprostol group): induction of labor by 25µg misoprostol oral tablet every 4 hours maximum200 µg.( Alfirevic Z et al., 2014)
2. nd group (Oxytocin group): oxytocin infusion according to ASUMH oxytocin protocol.

Syntocinon Mix: {if patient fit for induction} Put 3 international units "IU" oxytocin (3000mIU) +50ml of normal saline in syringe pump= (60mIU/ml).

Commence at 1ml/hour (1mIU/min) for 1/2 hour.

* If contractions inadequate +fetal monitor healthy 2 ml/hour for 1/2 hour.
* If contractions inadequate +fetal monitor healthy 4 ml/hour for 1/2 hour.
* If contractions inadequate +fetal monitor healthy 6 ml/hour for 1/2 hour.
* If contractions inadequate +fetal monitor healthy increase by 2ml/hr. for max. 27ml/hour.

At any point there's fetal or maternal distress (e.g. pathological FHR pattern, antepartum hemorrhage, etc.) the study intervention will be stopped, and the maternal/fetal condition will be managed by cesarean section.

5. Follow up: Continuous electronic fetal heart rate monitoring Maternal: vital data, uterine contractions, cervical changes (PV/4hours). Time to active phase (cervical dilatation: 6cm) will be noted, and then follow-up monitoring till delivery.

6. End point: Reaching maximum dose of drugs with failure of induction of labor in which another decision should be taken. Also, at any point there's fetal or maternal distress (e.g. pathological FHR pattern, antepartum hemorrhage, etc.) the study intervention will be stopped, and the maternal/fetal condition will be managed accordingly.

7. Data collection and recording case record form: The data will be collected in a case report form (age, parity, gestational age, blood pressure, bishop score on admission, time till active phase, induction to delivery interval, any side effects if present, mode of delivery, birth weight, neonatal intensive care unit (NICU) admission, Apgar score, hospital stay, maternal intensive care unit (ICU) admission.

Statistical analysis:

The collected data will be revised, coded, tabulated and introduced to a personal computer (PC) using Statistical package for Social Science (SPSS 20.0.1 for windows; SPSS Inc, Chicago, 2001). Quantitative variables will be expressed as mean and standard deviation (SD), or median and interquartile range (IQR) according to type of data. Qualitative variables are expressed as frequencies and percentages. Student t test and Mann Whitney test will be used to compare a continuous variable between two study groups. Chi square test will be used to examine the relationship between categorical variables. A P-value< 0.05 will be considered statistically significant.

Ethical and Safety Consideration:

This study will be done after approval of the ethical committee ,faculty of Medicine, Ain Shams University. Informed consent will be taken from all participants before recruitment in the study, and after explaining the purpose and procedures of the study. The investigator will obtain the written, signed informed consent of each subject prior to performing any study specific procedures on the subject. All data will be collected confidentially. At any point there's fetal or maternal distress (e.g. pathological FHR pattern, antepartum hemorrhage, etc.) the study intervention will be stopped, and the maternal/fetal condition will be managed accordingly.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age (36-42 weeks).
* Prelabor rupture of membranes within the last 24hours
* Vertex presentation

Exclusion Criteria:

1. History of medical diseases (HTN, diabetes milletus, systemic lupus erythematosus, cardiac, etc.).
2. Antepartum hemorrhage
3. Chorioamnionitis / prelabor rupture of membranes >24hours
4. Multiple pregnancy.
5. Abnormal fetal heart rate pattern upon admission
6. Intrauterine growth restriction
7. Fetal malpresentation.
8. Previous uterine scar.
9. Estimated fetal weight more than 4kg.
10. Patients already in labor
11. Contraindication for prostaglandin/oxytocin use (allergy,..)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2022-05-16 (Actual)

PRIMARY OUTCOMES:
vaginal delivery | immediately after the intervention
  rate of successful vaginal delivery

SECONDARY OUTCOMES:
induction to active phase time | during the intervention
  Time interval from starting induction till active phase (6cm dilatation)
Induction to delivery time | during the intervention
  Time interval from starting induction till delivery
Apgar score | The score is reported at 1 minute and 5 minutes after birth for all infants
  This scoring system provides a standardized assessment for infants after delivery. The Apgar score comprises five components: 1) color, 2) heart rate, 3) reflexes, 4) muscle tone, and 5) respiration, each of which is given a score of 0, 1, or 2.
NICU admission | within 24hours after birth
  number of newborns admitted to the neonatal intensive care unit
maternal side effects | during labour and within 24hours after birth
  number of participants with temperature >38 degree celsius

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed S Sweed, MD, Study Director — Professor; Gasser A Elbishry, MD, Study Chair — Professor
Locations (1):
- Ain Shams Maternity Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
planning to share the study protocol, and master-sheet.
Supporting Information: Study Protocol, Analytic Code
Time Frame: After study completion and for 6months later
Access Criteria: However, the repository is not decided upon yet

REFERENCES:
- [Background] Alfirevic Z, Aflaifel N, Weeks A. Oral misoprostol for induction of labour. Cochrane Database Syst Rev. 2014 Jun 13;2014(6):CD001338. doi: 10.1002/14651858.CD001338.pub3. PMID 24924489
- [Background] Zeteroglu S, Engin-Ustun Y, Ustun Y, Guvercinci M, Sahin G, Kamaci M. A prospective randomized study comparing misoprostol and oxytocin for premature rupture of membranes at term. J Matern Fetal Neonatal Med. 2006 May;19(5):283-7. doi: 10.1080/14767050600589807. PMID 16753768
- [Derived] Ahmed RHM, Sweed MSE, El-Bishry GA, Hassan RK. Oxytocin Versus Oral Misoprostol for Induction of Labor in Pregnant Women with Term Prelabor Rupture of Membranes: a Randomized Clinical Trial. Reprod Sci. 2023 Dec;30(12):3507-3514. doi: 10.1007/s43032-023-01290-0. Epub 2023 Jul 13. PMID 37442883